CLINICAL TRIAL: NCT00695500
Title: A Randomized, Double-blind, Placebo Controlled Trial (RCT) of Varenicline to Reduce Alcohol Consumption in Heavy Drinkers
Brief Title: Varenicline to Reduce Alcohol Consumption in Heavy Drinkers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vijay Ramchandani, Ph.D. (NIH)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Vijay Ramchandani, Ph.D., Clinical Investigator and Chief, Section on Human Psychopharmacology, National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080137; 08-AA-0137 (Other: NIH Office of Protocol Services)
Record Dates: First submitted 2008-06-11; First posted 2008-06-12 (Estimated); Results first posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Alcohol Drinking
Keywords: Varenicline; Alcohol; Alcohol Use
MeSH Terms: conditions — Alcohol Drinking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Experimental): Varenicline tablets, 2 mg per day for 3 weeks
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Placebo tablets, 0 mg per day for 3 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline tablets, 2 mg per day for 3 weeks
  Arms: Varenicline
Drug: Placebo — Placebo tablets, 0 mg per day for 3 weeks
  Arms: Placebo

SUMMARY:
This study will determine whether varenicline, a drug that acts on the brain's nicotine receptors and is used to help smokers stop smoking, will have an impact on alcohol self-administration.

People between 24 and 60 years of age who regularly consume alcoholic drinks (more than 15 drinks per week for women, and more than 20 drinks per week for men) may be eligible for this study. The study requires five outpatient visits and one overnight hospital admission at the NIH Clinical Center.

Participants undergo the following procedures:

Visit 1 (outpatient: 4-5 hours)

* Standard assessments, including vital signs measurements, breathalyzer test, blood and urine tests (including pregnancy test for females), questionnaires about mood, symptoms, alcohol use and smoking, if applicable
* Questionnaires about medical and psychological status
* Health assessment and assessment of alcohol drinking behavior

Visit 2 (outpatient: 8 hours)

* Standard assessments (see above)
* Computer-Assisted Self-infusion of Ethanol (CASE) session: Subjects will receive a priming intravenous infusion of alcohol. After 25 min, they will be allowed to give themselves additional exposures of alcohol over a period of 2 hours by pressing a button on a computer that controls the infusion pump.

Visit 3 (outpatient: 2 hours)

-Standard assessments

Visit 4 (outpatient: 8 hours)

* Standard assessments
* Brain functional magnetic resonance imaging scan (MRI). This test uses a magnetic field and radio waves to produce images of the brain. The patient lies on a table that can slide in and out of the scanner, wearing earplugs to muffle loud sounds that occur during the scanning process. Initial pictures are taken of the brain's structure and additional scans measure brain activity while the subject performs simple tasks.
* Alcohol Infusion. Subjects receive an intravenous infusion of alcohol while in the MRI scanner to measure the brain s response to alcohol.

Visit 5 (overnight)

* Standard assessments
* Repeat CASE session
* Interview about the subject's experiences participating in the protocol, including any symptoms and urges to drink

Visit 6 (outpatient)

* Standard assessments (without blood tests)
* Interview about participation in the study

Telephone follow-up

After 3 weeks, subjects are called to check on their symptoms and gather information on their drinking and, if applicable, smoking.

DETAILED DESCRIPTION:
Objective:

Considerable clinical and experimental evidence in humans and animal models links nicotine use with heavy alcohol consumption. Varenicline, an alpha4beta2 (nicotinic) acetylcholine receptor (nAchR) partial agonist, is an oral medication approved by the FDA (2006) for smoking cessation. Recently, it has been shown to reduce alcohol consumption in a rodent model of alcohol dependence. In the present short-term experimental study, it will be assessed primarily for its ability to reduce alcohol self-administration in heavy drinkers. Secondarily, its effects on alcohol urges (cravings), as well as smoking parameters will be measured. In addition, effects of varenicline on incentive motivation for alcohol and the underlying brain reward system activation, as well as on activation of brain reward systems in response to intravenously administered alcohol will be measured.

Study Population:

Fifty healthy, adults (smokers and non-smokers), age 21 to 60 years, will be studied. Individuals must drink alcohol regularly at a heavy level, on average greater than 20 drinks per week for men, and greater than 15 drinks per week for women, and not be seeking help for alcohol-related problems.

Design:

Following protocol screening and medical evaluation, qualified subjects will undergo an initial ( pre-study drug ) intravenous alcohol self-administration session (hereafter, called computer-assisted self-infusion of ethanol, or CASE). Following this, subjects will be randomized to varenicline or placebo. Subjects will be clinically evaluated on three occasions while on study drug: once after one week of study medication; again, prior to the fMRI; and again, at the end of treatment, when they undergo the second ( on-study drug ) CASE session. Between days 13 and 21, all subjects will be scheduled to undergo functional magnetic resonance imaging (fMRI) of the brain while performing a task designed to evaluate the incentive salience for alcohol cues as well as the pharmacological effects of alcohol. Thereafter, all subjects will receive two courses of counseling for heavy drinking, using motivational enhancement techniques, aimed at enhancing their readiness for behavioral change and seeking treatment, if needed.

Outcome Measures:

The primary outcome will be the peak breath alcohol exposure achieved during the on-study drug CASE session. Secondary outcomes during the study drug phase will include measures of alcohol consumption, and urges to drink, as well as alcohol cravings and effects during the on-study drug CASE session. Additionally, fMRI BOLD responses in the ventral striatum, an area involved in brain reward circuitry and shown to be activated by acute IV alcohol administration as well as anticipation of working for reward will be measured. In smokers, cigarette use and quite rates as well as urges to smoke and nicotine withdrawal will also be measured. Safety and tolerability will be followed during the course of taking study drug with symptom checklists, profiles of mood and anxiety and by clinical interview. Serum varenicline concentrations will also be measured to assess compliance and control for potential pharmacokinetic variation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 21 to 60 years of age.
* In good health.
* Drink a weekly average of 15 and 20 standard alcoholic drinks (12 gm ethanol/beverage), respectively, for women and men.
* Have a working phone number.

EXCLUSION CRITERIA:

* Currently seeking help for an alcohol problem.
* Subjects with clinically significant alcohol withdrawal.
* More than thirty days of abstinence from alcohol in the ninety days prior to enrollment.
* A positive breath alcohol concentration (BrAC) at the first visit
* A history of major alcohol-related complications at any time, such as pancreatitis.
* Any serious cardiovascular condition or high risk factors, evidenced by any of the following:

  * Current or past diagnosis of coronary artery disease (such as ischemia, angina, congestive heart failure, myocardial infarction) or peripheral arterial disease;
  * Current or past diagnosis of diabetes, or casual glucose level > 200 mg/dl;
  * Elevated blood pressure (above 160/100) at screening,
  * Elevated lipid levels: LDL > 160 mg/dL, HDL < 40 mg/dL for males or < 45 mg/dL for females;
  * Clinically significant ECG abnormalities or unstable arrhythmias.
  * Contraindication(s) to take the study medication as listed in the package insert.
* Contraindication(s) to take the study medication as listed in the package insert.
* Psychiatric problems requiring clinical attention: a current or past diagnosis of major depression, panic disorder, eating disorders, post traumatic stress disorder, schizophrenia, bipolar disorder, or obsessive compulsive disorder. Individuals who report lifetime (past or current) history of suicidal ideation, suicide attempts or self injury.
* Recent (within the last two months) or regular use of illicit or non-prescribed psycho-active substances such as opiates, benzodiazepines, cocaine, PCP, methamphetamines/other psychostimulants or marijuana.
* Psycho-social instability (e.g. no fixed address, no reliable secondary person to contact in case of an emergency).
* Women who are lactating, are trying to become pregnant or who are not willing to practice safe and effective birth control.
* Moderate-to-severe renal impairment defined as estimated or measured creatinine clearance less than 30 mL/min.
* Use of bupropion or nicotine replacement therapy within 90 days of the protocol, inhibitors/substrates for renal cationic transporters, or medications contraindicated with ethanol.
* Exclusion criteria for MRI scanning, including metal in body (such as implants, pacemaker, prostheses, shrapnel, irremovable piercing), left-handedness, and claustrophobia.
* A history of violence or aggression, assessed as part of the clinical interview at screening visit.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-06; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijay A Ramchandani, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lachin JM, Matts JP, Wei LJ. Randomization in clinical trials: conclusions and recommendations. Control Clin Trials. 1988 Dec;9(4):365-74. doi: 10.1016/0197-2456(88)90049-9. PMID 3203526
- [Background] Wei LJ, Lachin JM. Properties of the urn randomization in clinical trials. Control Clin Trials. 1988 Dec;9(4):345-64. doi: 10.1016/0197-2456(88)90048-7. PMID 3203525
- [Background] Falk DE, Yi HY, Hiller-Sturmhofel S. An epidemiologic analysis of co-occurring alcohol and tobacco use and disorders: findings from the National Epidemiologic Survey on Alcohol and Related Conditions. Alcohol Res Health. 2006;29(3):162-71. PMID 17373404
- [Derived] Gowin JL, Vatsalya V, Westman JG, Schwandt ML, Bartlett S, Heilig M, Momenan R, Ramchandani VA. The Effect of Varenicline on the Neural Processing of Fearful Faces and the Subjective Effects of Alcohol in Heavy Drinkers. Alcohol Clin Exp Res. 2016 May;40(5):979-87. doi: 10.1111/acer.13046. Epub 2016 Apr 8. PMID 27062270

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants were enrolled (consented) but withdrew prior to group assignment.
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 24 | 22
Completed | 21 | 17
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 22 | 21 | 43
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 23 | 21 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 14 | 9 | 23
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption
Description: Peak Breath Alcohol Concentration during IV alcohol self-administration
Time Frame: 2.5 hr session following 3 weeks of treatment
Population: sample that completed the assessment
Measure: Mean (Standard Error); unit: mg/%
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 16 | 12
mg/% | 92.0 (11.6) | 77.3 (13.5)

2. Secondary Outcome: Alcohol Urges
Description: Peak Alcohol Urge Questionnaire Score during IV alcohol self-administration. Scale: Alcohol Urge Questionnaire. Contains 8 items, each item scored on a likert scale from 1 to 7.
  Range: Total scores range between 8 and 64. Higher scores indicate higher urges for alcohol.
Time Frame: 2.5 hr session following 3 weeks of treatment
Population: sample that completed the assessment
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 16 | 12
Units on a scale | 23.65 (2.74) | 26.82 (3.70)

3. Other Pre Specified Outcome: BOLD Response to Alcohol Cue
Description: Percent BOLD signal change during Alcohol Food Incentive Delay Task (Alcohol - Neutral)
Time Frame: fMRI session following 2 weeks of treatment
Population: sample that completed the assessment
Measure: Mean (Standard Error); unit: Percent Signal Change
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 16 | 12
Percent Signal Change | -0.021 (0.051) | 0.194 (0.080)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 21/24 | 18/22
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=24) | Placebo (N=22)
Chest pain - cardiac (Cardiac disorders) | 4 | 1
Palpitations (Cardiac disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 7 | 6
Diarrhea (Gastrointestinal disorders) | 6 | 3
Flatulence (Gastrointestinal disorders) | 10 | 5
Nausea (Gastrointestinal disorders) | 14 | 6
Stomach pain (Gastrointestinal disorders) | 6 | 4
Irritability (General disorders) | 6 | 4
Anorexia (Metabolism and nutrition disorders) | 6 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 6
Headache (Nervous system disorders) | 11 | 8
Lethargy (Nervous system disorders) | 13 | 11
Memory impairment (Nervous system disorders) | 11 | 9
Somnolence (Nervous system disorders) | 7 | 6
Agitation (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 8 | 7
Psychiatric disorders - Other, specify (Psychiatric disorders) | 17 | 12
Uterine pain (Reproductive system and breast disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2

LIMITATIONS AND CAVEATS:
The IV alcohol self-administration method may have shown ceiling effects limiting the interpretation of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes